CLINICAL TRIAL: NCT00462670
Title: A Double-blind, Placebo-controlled Study of OPC-41061 in the Treatment of Cardiac Edema (Congestive Heart Failure)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-06-002
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2013-12

CONDITIONS: Edema, Cardiac
Keywords: Cardiac edema; OPC-41061; Vasopressin antagonist
MeSH Terms: conditions — Edema, Cardiac | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): 0mg
  Interventions: Drug: OPC-41061(Tolvaptan)
- 2 (Experimental): 15mg OPC-41061
  Interventions: Drug: OPC-41061(Tolvaptan)

INTERVENTIONS:
Drug: OPC-41061(Tolvaptan) — 0, 15mg of OPC-41061 per day for 7days p.o. administration

SUMMARY:
To evaluate the efficacy and safety of 7-day repeated oral administration of OPC-41061 15 mg or placebo in congestive heart failure (CHF) patients with extracellular volume expansion despite the use of a conventional diuretic.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects receiving one of the following diuretic treatments (including subjects scheduled to start treatment during the run-in observation period, 1)A loop diuretic at a daily dosage equivalent to 40 mg or more of furosemide, 2)Concomitant administration of a loop diuretic and a thiazide diuretic (at any doses), 3)Concomitant administration of a loop diuretic and an anti-aldosterone drug (at any doses)
2. CHF patients with lower limb edema, jugular venous distention, or pulmonary congestion due to extracellular volume expansion Patients with pulmonary congestion can be enrolled if pulmonary congestion is confirmed on chest x-ray taken within 14 days prior to the screening examination.
3. Male or female subjects age 20 or older and younger than 85 (at time of informed consent)
4. Subjects who are able to stay at the study site from the day before the start of the run-in observation period until completion of postdosing examination 2 (7 to 10 days after final study drug administration)
5. Subjects capable of giving informed consent to participate in the study of their own free will

Exclusion Criteria:

1. Subjects with acute heart failure
2. Subjects with an assisted circulation device
3. Subjects with any of the following complications or symptoms: (1)Suspected decrease in circulatory blood flow, (2)Hypertrophic cardiomyopathy (other than dilated phase), (3)Cardiac valve disease with significant heart valve stenosis, (4)Hepatic coma
4. Subjects who develop acute myocardial infarction within 30 days prior to the screening examination
5. Subjects with a definite diagnosis of active myocarditis or amyloid cardiomyopathy
6. Subjects with any of the following complications or symptoms: (1)Diabetes mellitus with poorly controlled blood glucose, (2)Anuria, (3)Urination impaired due to urinary tract stricture, urinary calculus, tumor in urinary tract, or other cause
7. Subjects with a history of any of the following diseases: (1)Sustained ventricular tachycardia or ventricular fibrillation within 30 days prior to the screening examination in patients without an implanted defibrillator, (2)Cerebrovascular disorder within 6 months prior to the screening examination (other than asymptomatic cerebral infarction), (3)Hypersensitivity or idiosyncratic reaction to benzazepine derivatives such as mozavaptan hydrochloride or benazepril hydrochloride.
8. Subjects who are obese [body mass index (BMI, body weight (kg)/height (m)2 exceeding 35]
9. Patients with supine systolic blood pressure exceeding 90 mmHg
10. Subjects with any of following abnormal laboratory values: (1)Total bilirubin exceeding 3.0 mg/dL, (2)serum creatinine exceeding 3.0 mg/dL, (3)serum sodium exceeding 147 mEq/L, (4)serum potassium exceeding 5.5 mEq/L
11. Patients who are unable to take oral medication
12. Female subjects who are pregnant, possibly pregnant, or lactating, or who plan to become pregnant
13. Subjects who received any investigational drug other than OPC-41061 within 30 days prior to the screening examination
14. Subjects who previously participated in this or any other study of OPC-41061 and received OPC-41061
15. Subjects otherwise judged by the investigator or subinvestigator to be inappropriate for inclusion in the study

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Division of New Product Evaluation and Development
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 0mg
  OPC-41061(Tolvaptan) : 0, 15mg of OPC-41061 per day for 7days p.o. administration
- OPC-41061 15mg: 15mg OPC-41061
  OPC-41061(Tolvaptan) : 0, 15mg of OPC-41061 per day for 7days p.o. administration
Period: Overall Study
Arm/Group | Placebo | OPC-41061 15mg
Started | 57 | 53
Completed | 52 | 46
Not Completed | 5 | 7
Not completed — Adverse Event | 3 | 5
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Resolution of signs and symptoms | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 0 mg of OPC-41061 per day for 7days p.o. administration
- OPC-41061: 15mg of OPC-41061 per day for 7days p.o. administration
- Total: Total of all reporting groups
Arm/Group | Placebo | OPC-41061 | Total
Number analyzed (Participants) | 57 | 53 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 12 | 31
  >=65 years | 38 | 41 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (10.9) | 71.3 (10.6) | 71.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 39 | 35 | 74
Region of Enrollment [Number; unit: participants]
  Japan | 57 | 53 | 110

OUTCOME MEASURES:

1. Primary Outcome: Body Weight (Amount of Change)
Description: Change in body weight from baseline at the time of final trial drug administration
Time Frame: baseline, Day 7 or at the time of final trial drug administration
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Placebo | OPC-41061 15mg
Number analyzed (Participants) | 57 | 53
Kg | -0.45 (0.93) | -1.54 (1.61)
Statistical Analysis 1: Comparison: Placebo vs OPC-41061 15mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -1.09, 95% CI 2-sided [-1.58 to -0.60], Standard Error of Mean 0.25

2. Secondary Outcome: Body Weight (Percent Change)
Description: Percent change in body weight from baseline at the time of final trial drug administration
Time Frame: baseline, Day 7 or at the time of final trial drug administration
Measure: Mean (Standard Deviation); unit: percentage of body weight (Kg)
Arm/Group | Placebo | OPC-41061 15mg
Number analyzed (Participants) | 57 | 53
percentage of body weight (Kg) | -0.77 (1.65) | -2.50 (2.55)
Statistical Analysis 1: Comparison: Placebo vs OPC-41061 15mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -1.73, 95% CI 2-sided [-2.54 to -0.92], Standard Error of Mean 0.45

ADVERSE EVENTS:
Time Frame: 7 days
Groups:
- OPC-41061 15mg: 15 mg of OPC-41061 per day for 7days p.o. administration
Arm/Group | Placebo | OPC-41061 15mg
Serious Adverse Events (participants affected / at risk) | 7/57 | 2/53
Other Adverse Events (participants affected / at risk) | 31/57 | 28/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | OPC-41061 15mg (N=53)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | OPC-41061 15mg (N=53)
Ventricular Extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 9 (10)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Face Oedema (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Thirst (General disorders) | 1 (1) | 9 (9)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Blood Creatinine Increased (Investigations) | 7 (7) | 4 (4)
Blood Potassium Increased (Investigations) | 4 (4) | 3 (3)
Blood Urea Increased (Investigations) | 10 (10) | 5 (5)
Blood Uric Acid Increased (Investigations) | 3 (3) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No